CLINICAL TRIAL: NCT07363018
Title: Efficacy of a Non-Invasive Endometrial Receptivity Prediction Model Based on Peripheral Blood miRNA Signatures During the Peri-Implantation Period in Improving IVF Outcomes in Patients With Unexplained Recurrent Implantation Failure: A Prospective, Single-Blind, Two-Arm, Parallel Randomized Controlled Trial
Brief Title: Efficacy of a Non-Invasive Endometrial Receptivity Prediction Model Based on Peripheral Blood miRNA Signatures During the Peri-Implantation Period in Improving IVF Outcomes in Patients With Unexplained RIF
Acronym: RIF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20251123
Record Dates: First submitted 2025-12-28; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Implantation Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Embryo Transfer Group (Experimental)
  Interventions: Diagnostic Test: Non-invasive endometrial receptivity prediction model guides personalized embryo transfer for patients with recurrent implantation failure (RIF).
- Standard Embryo Transfer Group (No Intervention)

INTERVENTIONS:
Diagnostic Test: Non-invasive endometrial receptivity prediction model guides personalized embryo transfer for patients with recurrent implantation failure (RIF). — Participants will undergo personalized embryo transfer based on the detection results of the window of implantation (WOI) via peripheral blood miRNA analysis. For subjects whose WOI results indicate that Day 5 (D5) is non-receptive, the embryo transfer timing will be appropriately advanced or delayed by 24 or 48 hours relative to the standard time. For subjects whose WOI results indicate that D5 is receptive, embryo transfer will be performed at the standard time (the fifth day after ovulation).
  Arms: Individualized Embryo Transfer Group

SUMMARY:
The goal of this clinical trial aims to investigate whether a non-invasive implantation window prediction model, constructed based on characteristic changes in peripheral blood miRNAs during the peri-implantation period, can improve pregnancy outcomes in patients with unexplained recurrent implantation failure undergoing frozen embryo transfer. Researchers will compare the clinical pregnancy outcomes between individualized embryo transfer guided by implantation window results and conventional embryo transfer, to observe whether implantation window-guided individualized embryo transfer can improve the clinical efficacy for patients with recurrent implantation failure (RIF). Participants will complete implantation window testing as required by the study protocol, undergo randomization and blinding, and proceed with embryo transfer according to their assigned group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unexplained recurrent implantation failure (RIF) meeting the diagnostic criteria for RIF: adult women under 40 years old who have failed to achieve clinical pregnancy after 3 embryo transfer cycles; or after transferring at least 3 high-quality embryos.

   Definition of high-quality embryos: Day 3 embryos (with a cell count ≥7 and fragmentation rate <10%) and blastocysts (≥3BB).
2. Female BMI: 18.5-25 kg/m².
3. Endometrial thickness ≥7 mm during the embryo transfer cycle.
4. Women planning to undergo frozen-thawed embryo transfer (FET) of blastocysts following in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI).
5. Signed informed consent form.

Exclusion Criteria:

1. Known causes of embryo implantation failure, such as infections, reproductive tract malformations, uterine cavity factors, adenomyosis or endometriosis, autoimmune system diseases (diagnosed by immunology department), hydrosalpinx, etc.
2. Couples with chromosomal abnormalities (excluding chromosomal polymorphisms) or familial genetic disorders in either or both partners.
3. Women with a history of recurrent miscarriage.
4. Women with contraindications to pregnancy or assisted reproductive technology.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 546 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Implantation rate per embryo transferred, assessed by counting gestational sacs on ultrasound. | From the day of embryo transfer until the completion of the first ultrasound assessment (typically at 35 days ± 7 days after transfer).
  Implantation rate is defined as the number of gestational sacs observed on ultrasound divided by the total number of embryos transferred. It will be expressed as a percentage: (Total number of gestational sacs / Total number of embryos transferred) × 100%. Assessment will occur approximately 35 days after embryo transfer.

SECONDARY OUTCOMES:
Proportion of patients with abnormal endometrial receptivity, as assessed by dynamic changes in peripheral blood microRNA levels 5 days after ovulation. | From the day of ovulation trigger until the completion of microRNA sample collection and analysis (within 5 to 7 days post-trigger).
  Endometrial receptivity will be assessed via the dynamic changes in specific microRNA expression profiles in peripheral blood, measured 5 days after ovulation (day of trigger). The "abnormal receptivity" (non-receptive) status is defined as a microRNA profile falling outside the established reference range for the receptive phase. The proportion will be calculated as: (Number of patients with a non-receptive microRNA profile / Total number of patients measured) × 100%.
Clinical pregnancy rate per embryo transfer, confirmed by ultrasound visualization of gestational sac and fetal heartbeat. | From the day of embryo transfer until the confirmation of clinical pregnancy by ultrasound (assessed at approximately 35 days ± 7 days after embryo transfer).
  Clinical pregnancy is defined as the presence of at least one intrauterine gestational sac with detectable fetal cardiac activity on transvaginal ultrasound. The rate will be calculated as: (Number of cycles achieving clinical pregnancy / Number of cycles with embryo transfer) × 100%.
Ongoing Pregnancy Rate per embryo transfer, confirmed by ultrasound after 12 weeks of gestation. | From the day of embryo transfer until the confirmation of fetal viability at or after 12 weeks of gestation (typically up to 14 weeks of gestation).
  Ongoing pregnancy is defined as an intrauterine pregnancy with confirmed fetal viability beyond 12 weeks of gestation (i.e., after the first trimester). The rate will be calculated as the number of cycles achieving an ongoing pregnancy divided by the number of cycles with embryo transfer, expressed as a percentage: (Number of ongoing pregnancies / Number of embryo transfer cycles) × 100%. Fetal viability will be assessed via transvaginal or abdominal ultrasound, demonstrating the presence of fetal cardiac activity.